CLINICAL TRIAL: NCT05614531
Title: A Multicenter, Nonrandomized, Open-label,Dose Escalation Clinical Trial to Assess the Safety and Efficacy of EXG001 307 After Intravenous Injection in Patients with Spinal Muscular Atrophy Type 1
Brief Title: Clinical Trial to Assess the Safety and Efficacy of EXG001-307 in Patients with Spinal Muscular Atrophy Type 1
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXG001-307-102; 2022LP00989 (Other: National medical Products Administration of China)
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spinal Muscular Atrophy Type I
Keywords: SMA，SMA1
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation- Cohort 1 (Experimental): dose 1 of EXG001-307 delivered one-time through a venous catheter inserted into a peripheral vein (n=3~6)
  Interventions: Genetic: EXG001-307 injection
- Dose escalation-Cohort 2 (Experimental): dose 2 of EXG001-307 delivered one-time through a venous catheter inserted into a peripheral vein (n=6~12)
  Interventions: Genetic: EXG001-307 injection
- Dose escalation-Cohort 3 (Experimental): dose 3 of EXG001-307 delivered one-time through a venous catheter inserted into a peripheral vein (n=3~6)
  Interventions: Genetic: EXG001-307 injection

INTERVENTIONS:
Genetic: EXG001-307 injection — non-replicating, rAAV vector based on AAV9 containing cDNA encoding the human SMN protein.

SUMMARY:
The purpose of this trial is to evaluate safety and efficacy of intravenous delivery of EXG001-307 as a treatment of spinal muscular atrophy Type 1 (SMN1).

DETAILED DESCRIPTION:
The study will evaluate safety and efficacy of gene therapy in spinal muscular atrophy Type 1 (SMA1) patients. SMA is caused by low levels of the survival motor neuron (SMN) protein, and affects all muscles in the body. There is no effective treatment for SMA and current drug therapy has been unsuccessful in stabilizing or reversing this disease. Only supportive care is currently possible.

Open-label, dose-escalation clinical trial of EXG001-307 injected intravenously through a peripheral limb vein. Short-term safety will be evaluated over a 1.5 year period. Patients will be tested at baseline and return for follow up visits on days 14, 21, 30, followed by once every month through 12 months post dose, and then every three months through a year and a half post infusion. Unscheduled visits may occur if the PI determines that they are necessary.

The primary analysis for efficacy will be assessed when all patients reach 18 months of age (a database lock will be performed at the time point at which all patients reach 18 months of age). A follow-up safety analysis will be completed at the time point at which the last patient reaches 18 months of age after post-dose.

Upon completion of the 1.5-year study period, patients will be monitored annually as per standard of care for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. SMA was diagnosed by a bilaterally allelic SMN1 mutation (deletion or point mutation) gene with 2 copies of the SMN2 gene.
2. On the day of dosing, the subject ' s age did not exceed postnatal Day 180.
3. The clinical history and signs were consistent with type 1 SMA manifestations, i.e. hypotonia, delayed motor function development, poor head control, round shoulder posture, and joint hypermobility.
4. The subject's legal guardian understands the purpose, possible risks and interests of the study, agrees to participate in the study, completes all study procedures, tests and visits, and voluntarily signs the informed consent form.
5. During the study, the subject's legal guardian was willing to perform standard treatment requirements such as nasogastric feeding, noninvasive mechanical ventilation, and expectoration machine as recommended by the investigator.

Exclusion Criteria:

1. Gestational age at birth was less than 35 weeks (245 days).
2. At screening, the subject had an oxygen saturation < 96% while awake or sleeping and did not receive any supplemental oxygen or respiratory support.
3. Requirement of invasive ventilation or tracheotomy, or current use of noninvasive ventilatory support for an average of ≥ 16 hours/day.
4. Weighed below the 3rd percentile by age according to the WHO Child Growth Criteria (WHO 2009).
5. Before administration, if the subject has not received or delayed vaccination according to the current month-old national vaccination plan, it will significantly affect the safety of the subject as assessed by the investigator and the medical manager of the project team;
6. Active viral infections (including HIV, COVID-19, hepatitis B or C seropositivity, torch virus, Epstein-Barr virus, and syphilis).
7. Serious non-respiratory disease within 2 weeks prior to screening.
8. Upper respiratory tract infection or lower respiratory tract infection within 4 weeks prior to screening.
9. Current presence of other severe infections or diseases.
10. Known cardiac disease or ECG abnormalities that are clinically significant.
11. Known hypersensitivity to prednisolone, other glucocorticoids, or its excipients.
12. Immunosuppressive therapy (eg, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, rituximab) other than protocol-required prophylaxis within 3 months prior to dosing.
13. Immunomodulatory drugs (eg, thymosin, interferon, etc.) are being used to treat myopathy, neuritis, diabetes mellitus (eg, immunosuppressants, glucocorticoids, insulin).
14. Anti-AAV9 antibody titer > 1: 50 (as determined by ECL). If the potential subject has an anti-AAV9 antibody titer > 1: 50, it can be retested during the screening period. If the anti-AAV9 antibody titer is ≤ 1: 50 at the retest, the subject may continue to participate in the screening.
15. Clinically significant abnormal laboratory values (GGT, ALT, and AST > 2.5 × ULN, bilirubin ≥ 3.0 mg/dL, creatinine ≥ 1.0 mg/dL, hemoglobin < 8 or > 18 g/dL; white blood cell count > 20,000/cm3; platelet count < 100,000/cm3).
16. Prior use of other SMA therapeutic agents (e.g., nosinasenat, rispolam, and Zolgensma, etc.) or participated in clinical studies with other SMA therapeutic agents (including but not limited to the above 3 drugs).
17. Major surgery is expected during study treatment.
18. Other circumstances that, in the judgment of the investigator, are not suitable for participation in this study.

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of EXG001-307 following a single intravenous infusion | During each visit
  including type and incidence of AE, SAE, AESI, vital signs, physical/neurological examination, immunogenicity, virology, injection/infusion site reactions, 12-lead electrocardiogram, and safety laboratory results recorded

SECONDARY OUTCOMES:
Patients number who survival at 14 month of age | up to 14 month of age
  survival at 14 months of age was defined as the number of participants who did not die, did not require permanent ventilation (defined as absence of acute reversible disease [excluding perioperative ventilation], requiring tracheotomy or respiratory assistance with non-invasive ventilation support for ≥16 hours per day for ≥14 consecutive days) and did not withdraw from the study by 14 months of age.
Number of patients who were able to sit unsupported for ≥30 seconds | From Day 1 up to 18 Months of Age Visit
  According to the Bailey Scale of Infant and Child Development Version 3 (BSID-III) ,sit unsupported as a participant who sits up straight with head erect for at least 30 seconds; participant does not use arms or hands to balance body or support position, evaluation procedure will confirmed by video recording

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Children'S Hospital Zhejiang University of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song C, Wang Q, Zhu P, Li J, Dai L, Hu W, Yang W, Zhang R, Wang D, Li Z, Chen S, Wang L, Ye G, Wu Z. Efficacy and preliminary safety assessment of EXG001-307 AAV gene therapy for spinal muscular atrophy. Mol Ther Methods Clin Dev. 2025 Apr 18;33(2):101475. doi: 10.1016/j.omtm.2025.101475. eCollection 2025 Jun 12. PMID 40458203